

# SAFE Spaces Staff Participation Consent Form Brief Summary

You have been invited to take part in a study to understand how the SAFE Spaces intervention program of staff-focused wellness supports and skill development opportunities can create safer and healthier environments for staff and youth in residential facilities. If you agree to participate in this study, you will be asked to do the following:

- 1. If your site is randomly assigned to receive the SAFE Spaces program, you will be offered flexible wellness supports and skill development tools.
- 2. Regardless of whether your site is assigned the SAFE Spaces program, you will be invited to answer survey questions every 6 months to receive a gift card.
  - a. The gift card for the first survey is \$20. The gift card for the 6-month survey is \$40. The gift cards for the 12-month, 18-month, and 24-month surveys are \$50.
  - b. You will also be entered into a raffle to win a \$1,000 prize for every survey you complete. Raffle winners will be drawn about every 6 months. There is about a 1 in 150 chance that you will win a raffle.

Each survey should take about 60 minutes to complete. While there are no known risks associated with your participation in this research, you may find some questions to be sensitive in nature, and you may skip questions or quit participating at any point. By answering survey items, you will help us understand how providing wellness skills and supports to staff creates safer and healthier environments for staff and young people in CTH.

The purpose of this study is to evaluate the safety and effectiveness of the SAFE Spaces program. You should know that if you are assigned to a facility receiving the program, we cannot guarantee that it will be as effective as the standard training you receive.

Participation in this study is voluntary. You may refuse to participate or withdraw at any time without penalty. Please read the rest of this permission form for more information about the study.

I want to begin by thanking you for letting us invite you to be a part of the SAFE Spaces project. This form will describe the research study and asks if you would like to participate. Dr. Shabnam Javdani and Dr. Erin Godfrey at the Steinhardt School of Culture, Education, and Human Development at New York University are the principal investigators of the research project, which is funded by the National Institutes of Mental Health (NIMH). Please feel free to ask any questions that you may have at any point. If you have any questions later, you can contact Dr. Javdani at 212-992-9739, <a href="mailto:shabnam.javdani@nyu.edu">shabnam.javdani@nyu.edu</a> or Dr. Godfrey at 212-998-5396, <a href="mailto:erin.godfrey@nyu.edu">erin.godfrey@nyu.edu</a>.

Why am I being invited to take part in this research study?



You are being invited to participate in a research study conducted by New York University because you work with or on behalf of youth in residential facilities. The study is called SAFE Spaces. As part of the study, we are providing wellness supports to staff that work with kids who live in residential facilities. We want to know how these supports help create safer and healthier environments for staff and young people.

Because of this, some facilities will get offered the SAFE Spaces program, and some will not until the study period is over. Whether a facility is chosen to get the SAFE Spaces program is completely random, like flipping a coin. None of the other trainings, programs or services that are offered to staff in your facility will be impacted by which group your facility gets assigned to. It is very important to learn from the perspective of staff about whether the SAFE Spaces program works. For this reason, you will be invited to fill out surveys, regardless of whether your facility has been assigned to the SAFE Spaces program or not.

### Why is this research study being done?

We are doing this research study because we want to increase youth and staff safety and well-being in residential facilities, and one important way to do that is through supporting staff.

## What happens if I say "Yes, I want to be in this research study?"

If your facility has been randomly assigned to receive the SAFE Spaces program:

- You will be offered wellness supports and skill development opportunities through coach visits to your facility.
- You will be invited to complete surveys about every 6 months during the study period.
- Your participation in the wellness skills and supports and the surveys are separate: You can take advantage of the wellness skills and supports and not complete the surveys, or complete the surveys and not use the wellness skills and supports.
- Whether or not you decide to participate in the SAFE Spaces program will be kept confidential and not affect your employment status or performance evaluation in any way.

### If your site is randomly assigned not to receive the SAFE Spaces program:

• You will be invited to complete surveys about every 6 months during the study period.

### What happens if I say "No, I do not want to be in this research study?"

- If you do not want to participate in the research study, you will not be asked to answer survey questions.
- If your facility has been assigned to the SAFE Spaces program, you may choose to use those wellness skills and supports, even if you do not wish to answer survey questions as a part of the research study.
- You receive all your usual training opportunities outside of the SAFE spaces program and research study.
- Whether or not you decide to participate in the SAFE spaces research study will be kept confidential and not affect your employment status or performance evaluation in any way.



## What are the surveys?

You will be invited to complete surveys for the length of the study period which is about 2 years, or only for as long as you are working in a residential facility. Each survey should take about 60 minutes to complete.

- Starting now and every 6 months afterwards during the study period, you will be asked to complete a survey. You will receive a gift card for your time. The gift card for the first survey is \$20. The gift card for the 6-month survey is \$40. The gift cards for the 12-month, 18-month, and 24-month surveys are \$50 each.
- Each time you participate in a survey, you will be entered into a raffle to win a \$1000 prize. One raffle winner will be drawn about every six months. There is about a 1 in 150 chance that each participant will win a raffle each year.
  - i. The \$1000 raffle prize payment will be reported to the IRS as compensation. If you are a raffle winner, you will be issued a 1099 form and required to submit a W-9 form with your Social Security Number and home address.

Please note that participation is completely voluntary. You may refuse to participate or withdraw from the study at any time without penalty. You have the right to skip or not answer any questions you prefer not to answer. There are no right or wrong answers to survey questions. Nonparticipation or withdrawal will not be reported to anyone outside of the research team and will in no way affect your position status. Your name will only be removed from entry in the raffle that is due to happen after you withdraw participation.

#### What are the risks and benefits?

- Risk: Although every effort will be made to prevent it, you may find the sensitive nature of some of the questions upsetting. In this case, you may skip questions or quit participating at any time without penalty or explanation.
- Risk: Your responses will be kept confidential with the following exception: (1) If you share that there is risk of hurting yourself or (2) If you share that a child under the age of 18 is experiencing abuse, the team is required by law to report it to the appropriate authorities.
- Benefit: Participation in this study will help us to understand how the SAFE Spaces program works. Please note that we cannot guarantee that the SAFE Spaces staff training program will be more effective than the standard training you receive as a part of your position. However, by answering survey items, you will help us learn more about your experiences, which can help us understand if providing wellness skills and supports to staff creates safer and healthier environments for staff and young people in residential facilities and can inform the legal system about best practices.

#### How do we make sure our research records are confidential (private)?

- Your name and personal information will always be kept separate from your survey answers.
- Your survey answers, if they are on paper, will be kept stored in a locked cabinet in a locked room of the research laboratory, with the Principle Investigators and senior research staff being the only ones to have access to the keys.



- Electronic files will be kept on a secure server on secure computers. Only members of the research team will have access to this secure server.
- Identifiable information about you will not be shared.
- You are welcome to request copies of any of the forms you complete.
- The only time we might have to share what you say with others is if you provide information concerning the abuse or neglect of a child under the age of 18, and if we learn about serious risks of harm to oneself or others.
- Information not containing identifiers may be used in future research, shared with other researchers, or placed in a data repository without your additional consent.

A description of this clinical trial will be available on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a>, as required by U.S. Law. This website may include a summary of the results, but will never include information that can identify you. You can search this website at any time. This research is covered by a Certificate of Confidentiality from the National Institutes of Health. Researchers with this Certificate will not disclose or use information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or any other action, suit, or proceeding, even if there is a court subpoena. Exceptions include:

- A federal, state, or local law requires disclosure (such as information about suspicion of child abuse or neglect, suspicion of harm to yourself or others).
- Your explicit approval for the researchers to release your name and/or personally identifiable information.

#### **Further Information:**

If there is anything about the study or your participation that is unclear or that you do not understand, if you have any questions or wish to report a research-related problem, you may contact Dr. Javdani or Dr. Godfrey. For questions about your rights as a research participant, you may contact the University Committee on Activities Involving Human Subjects, New York University, 665 Broadway, Suite 804, New York, NY 10012 at 212-998-4808 or ask.humansubjects@nyu.edu.

| University, 665 Broadway, Suite 8 ask.humansubjects@nyu.edu. | 804, New York, NY 10012 at 212-998-4808 or |
|---|---|
| ********* | *************** |
| the information on this form and | signing below means that you have read and understand d that you agree to participate in the SAFE Spaces research im to use your answers on the questionnaires for research |
| I,(Print full name) | , have read all of the information above |
| responses for research purposes. | e. I agree to allow the SAFE Spaces research team to use my I had a chance to ask questions, I understand what this form ption to keep a copy of this consent form. |
| Staff signature | Date |



Do you give us permission to contact you for future opportunities to participate in research with our team?

- YES, I agree and give permission
- NO, I don't agree or give permission